CLINICAL TRIAL: NCT01631383
Title: Pharmacokinetic and Safety Evaluation of L-tetrahydropalmatine (l-THP) With Cocaine Exposure in People With a History of Cocaine Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, MPRC, Deanna L. Kelly, Pharm.D., BCPP, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00051290; 1DP1DA031401-01 (NIH)
Record Dates: First submitted 2012-06-18; First posted 2012-06-29 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Cocaine Use
Keywords: Cocaine Use

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- l-THP (Active Comparator)
  Interventions: Drug: l-THP (l-tetrahydropalmatine)

INTERVENTIONS:
Drug: l-THP (l-tetrahydropalmatine) — Subjects will arrive the first day (Day 1) for admission and morning l-THP dosing. The l-THP will be dosed as one capsule 30 mg twice daily (matching placebo or l-THP) (total 60 mg daily). Participants will receive 7 total l-THP doses: two doses on Day 1 (morning and evening), two doses on Day 2 (morning and evening), 2 doses on Day 3 (morning and evening) and one dose the morning of Day 4 (cocaine administration day).
  Other Names: l-tetrahydropalmatine
  Arms: l-THP
Drug: Placebo — Subjects will arrive the first day (Day 1) for admission and morning l-THP dosing. The l-THP will be dosed as one capsule 30 mg twice daily (matching placebo or l-THP) (total 60 mg daily). Participants will receive 7 total l-THP doses: two doses on Day 1 (morning and evening), two doses on Day 2 (morning and evening), 2 doses on Day 3 (morning and evening) and one dose the morning of Day 4 (cocaine administration day).
  Arms: Placebo

SUMMARY:
This study will test the safety and pharmacokinetic profile of l-THP with cocaine exposure in people who have a history of cocaine use. The subject will be admitted to the Brief Stay Unit (BSU), an inpatient facility at the Maryland Psychiatric Research Center, used for short term drug abuse or clinical trial studies. The participant will stay for 4 nights and 5 days. He/she will be randomized to either placebo or l-THP for three days. On the morning of Day 4, the subject will receive one cocaine dose (40 mg intranasal) and have testing for pharmacokinetic parameters for the following 10 hours. The subject will stay over one more night and will be discharged the following day. Approximately 40 subjects will be randomized to enroll the target sample of 30 (N=15 placebo, N=15 l-THP). In summary, each subject will come for a screening visit(s), then a 5-day, 4-night stay on a secure research unit. After cocaine administration day, the participant will stay overnight for one more day of observation and to permit substantial l-THP elimination from the body. The following morning we will get one additional blood specimen for l-THP (Day 5 at 24 hours after last dose (7:30 am); then the participant will be discharged. A visit with blood collection on Day 6 at 55 hours after last dose (2:30 pm) will be scheduled. A final follow-up visit will be scheduled 4-7 days after unit discharge to ensure no persisting side effects.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

Inclusion criteria:

1. men or non-pregnant/non-nursing women between the ages of 18 and 50 years old
2. self reported history of cocaine use (intranasal, IV or smoked) averaging at least twice monthly for at least one month over the prior year
3. self- reported use at least one use in the past six months of a cocaine dose equivalent to 40 mg intranasal or 15 mg smoked or intravenous, based on participant's best estimate of weight and/or street price of amount ingested and a
4. positive urine drug test for cocaine use at least once in past 1 year
5. HIV seronegative
6. hepatitis C seronegative
7. EKG without clinically significant abnormality
8. normal blood pressure (systolic: 90-140 mmHg; diastolic: 50-90 mmHg) and resting heart rate (60-90 bpm)
9. within 20% of ideal body weight, based on BJ Devine formula (1974) (men: 50 + 2.3 kg per inch over 5 feet, women: 45.5 + 2.3 kg per inch over 5 feet)
10. ability to adhere to the study restrictions and examination schedule
11. Women with reproductive potential must agree to the use of one of the following birth control methods (condom with spermicide, diaphragm, or intrauterine device) during the study and for 2 weeks after study conclusion.

Exclusion criteria:

1. participation in any investigational drug trial or clinical drug trial within 45 days before study entry
2. donation or loss of greater than one pint of blood within 60 days of study entry
3. history of clinically significant adverse reaction or hypersensitivity to any study drug,
4. inability to communicate or co-operate with the investigators
5. treatment-seeking for cocaine abuse/dependence
6. taking any concurrent prescription, over the counter medications, or dietary/nutritional/herbal supplement (such as St. John's wort or grapefruit juice, but not including standard vitamin or mineral supplements) within 14 days prior to initial dosing.
7. current clinically significant medical problems that might interfere with safe study participation. This includes pheochromocytoma, untreated hyperthyroidism, dehydration, fever, coronary artery disease, uncorrected congenital heart defect, seizures, electrolyte imbalance, uncontrolled diabetes mellitus, porphyria variegate, superventricular tachycardia, atrial fibrillation, cardiomyopathy, uncontrolled hypertension,.
8. Current Axis I psychiatric disorder (except nicotine dependence, cocaine abuse/dependence, or simple phobia). Nicotine does not alter physiologic response to cocaine (Kouri et al 2001)
9. Positive for illicit drugs other than cocaine or marijuana on urine drug screen
10. Score below 10/12 on the Evaluation to Sign Consent (ESC)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Peak heart rate after cocaine administration during treatment with l-THP or placebo. | -10 (min), 5, 20, 35, 50, 65, 80, 95, 2.5 (hr), 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9 10 hr
  Comparing the peak changes between the two groups accounting for the specified tolerance margin
Peak blood pressure after cocaine administration during treatment with l-THP or placebo | -10 (min), 5, 20, 35, 50, 65, 80, 95, 2.5 (hr), 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9 10 hr
  Comparing the peak changes between the two groups accounting for the specified tolerance margin
Peak cocaine plasma concentration after acute cocaine dose during treatment with l-THP | 0,1,20,30,40,50,60,70,80,90, 100, 110 (min), 2 (hr), 2.5, 3, 3.5, 4, 5, 6 hr
  Cmax and AUC will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L. Kelly, Pharm.D., BCPP, Principal Investigator — University of Maryland, College Park
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- See also: Maryland Psychiatric Research Center — http://www.mprc.umaryland.edu